CLINICAL TRIAL: NCT04764747
Title: Evaluating Effectiveness of Convalescent Plasma and Factors Influencing Therapeutic Outcome in Hospitalized Patients With COVID-19
Brief Title: Effectiveness of Convalescent Plasma in Hospitalized Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Kufa University (Other)
Responsible Party: Principal Investigator, Zainab Hadi Ibadi, Ms.Ph. Zainab Hadi Ibadi, Kufa University
Other Study IDs: CP in COVID-19 patients
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter retrospective cohort study from June to August 2020 on hospitalized COVID-19 patients admitted to Al-Hakeem and Al-Amal hospital in Al-Najaf Governorate, Iraq, in order to evaluating the effectiveness of plasma therapy in hospitalized patients with COVID-19 and analyzing factors that affect therapeutic outcome, either related to patients or related to donors.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is a contagious disease with high rate of fatality caused by severe acute respiratory syndrome coronavirus 2 (SARS-COV-2). In Wuhan, the capital of China's Hubei province, the disease was first detected in December 2019 and has since spread globally, resulting in the continuing 2019 and 2020 coronavirus pandemic. The World Health Organization (WHO) has proclaimed that on 30 January 2020, the outbreak will be a public health emergency of international concern and will be known as a pandemic on 11 March 2020. To date, no unique antiviral therapy or effective disease-containing vaccine exists. Therefore, it is an urgent need to look for an alternative strategy for COVID-19 treatment, especially among severe patients. For more than a century, convalescent plasma (CP) therapy, a classic adaptive immunotherapy, has been used to prevent and treat many infectious diseases. CP therapy has been successfully used in the treatment of severe acute respiratory syndrome (SARS), Middle east respiratory syndrome (MERS), and the 2009 H1N1 pandemic with adequate effectiveness and protection over the past two decades. For patients with serious or life-threatening COVID-19, the US Food and Drug Administration (FDA) recently approved the emerging use of convalescent plasma. While the use of convalescent plasma looks promising, there is still little evidence supporting its use in the treatment of COVID-19 and its use is therefore still investigational.

Also, there is lack of standardization and evidence-based rationale in donor eligibility requirements account for factors such as age, sex, weight, symptom course, antibody titer and it is association with clinical outcome. Additionally, recipient related factors including age, sex, weight, disease severity, time of CP use and concomitant treatment must be considered in prediction the response to CP therapy and this may help to explain the varied therapeutic effects of CP seen in a variety of studies. Considering the above-mentioned facts and high number of patients treated with CP in AL Najaf-Hakeem hospital and Amal hospital we designed this study to evaluate the effectiveness of CP therapy in hospitalized patients with COVID-19 and find patients and donor related factors to predicts the responders and not responders.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years old or older.
* COVID-19 confirmed by reverse transcriptase-polymerase chain reaction (RT-PCR).
* hospitalized adult patients with COVID-19.

Exclusion Criteria:

* Patients with history of alleragy to plasma transfusion.
* Patients with history of autoimmune disease or selective IgA deficiency.
* Patients with suspected coronavirus.
* Patients with incomplete data in his record.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients diagnosed with COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement | 14 days
  modified six-point ordinal scale of COVID-19
Find the prediction factors associated with good outcome of patients on CP therapy | 14 days
  Demographic data and clinical parameters of patients associated with positive therapeutic outcome for CP measured as number of patients discharge from hospital with complete recovery (negative PCR for COVID-19). The association determined by univariate and multivariate analysis
Time to negative PCR | 14 days
  number of days required for patients to be have negative PCR (free viral load)

SECONDARY OUTCOMES:
Mortality rate | 21 days
  number of deaths
Hospital stay time | 21 days
  duration of stay in hospital
Adverse effect of plasma therapy | 21 days
  to asses the frequency of adverse effect of convalescent plasma

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - Al-Amal Hospital, Najaf
  - Al-Hakeem Hospital, Najaf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chauhan S. Comprehensive review of coronavirus disease 2019 (COVID-19). Biomed J. 2020 Aug;43(4):334-340. doi: 10.1016/j.bj.2020.05.023. Epub 2020 Jun 1. PMID 32788071
- [Background] Li L, Zhang W, Hu Y, Tong X, Zheng S, Yang J, Kong Y, Ren L, Wei Q, Mei H, Hu C, Tao C, Yang R, Wang J, Yu Y, Guo Y, Wu X, Xu Z, Zeng L, Xiong N, Chen L, Wang J, Man N, Liu Y, Xu H, Deng E, Zhang X, Li C, Wang C, Su S, Zhang L, Wang J, Wu Y, Liu Z. Effect of Convalescent Plasma Therapy on Time to Clinical Improvement in Patients With Severe and Life-threatening COVID-19: A Randomized Clinical Trial. JAMA. 2020 Aug 4;324(5):460-470. doi: 10.1001/jama.2020.10044. PMID 32492084
- [Background] Duan K, Liu B, Li C, Zhang H, Yu T, Qu J, Zhou M, Chen L, Meng S, Hu Y, Peng C, Yuan M, Huang J, Wang Z, Yu J, Gao X, Wang D, Yu X, Li L, Zhang J, Wu X, Li B, Xu Y, Chen W, Peng Y, Hu Y, Lin L, Liu X, Huang S, Zhou Z, Zhang L, Wang Y, Zhang Z, Deng K, Xia Z, Gong Q, Zhang W, Zheng X, Liu Y, Yang H, Zhou D, Yu D, Hou J, Shi Z, Chen S, Chen Z, Zhang X, Yang X. Effectiveness of convalescent plasma therapy in severe COVID-19 patients. Proc Natl Acad Sci U S A. 2020 Apr 28;117(17):9490-9496. doi: 10.1073/pnas.2004168117. Epub 2020 Apr 6. PMID 32253318
- [Background] Farhat RM, Mousa MA, Daas EJ, Glassberg MK. Treatment of COVID-19: Perspective on Convalescent Plasma Transfusion. Front Med (Lausanne). 2020 Jul 28;7:435. doi: 10.3389/fmed.2020.00435. eCollection 2020. PMID 32850916